CLINICAL TRIAL: NCT03123302
Title: Our Anesthesia Experience During MRI Scan
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, İlker Onguc Aycan, department of anesthesiology and reanimation, Akdeniz University
Other Study IDs: MEDAH
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Epileptic Seizure; Intracranial Tumor; Intracranial Hypertension; Intracranial Aneurysm; Vertebra; Anomaly
Keywords: MRI scan, sedation, epilepsia
MeSH Terms: conditions — Seizures; Brain Neoplasms; Intracranial Hypertension; Intracranial Aneurysm; Congenital Abnormalities; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Epileptic patients who are sedated with a total dose of propofol 2 mg/kg and midazolam 0.1 mg/kg.
- Group 2: Epileptic patients who are sedated with a total dose of pentothal 4 mg/kg and midazolam 0.1 mg/kg.
- Group 3: Non-epileptic patients who are sedated with a total dose of propofol 1 mg/kg and ketamine 1 mg/kg.
- Group 4: Non-epileptic patients who are sedated with a total dose of midazolame 0.1 mg/kg and ketamine 1 mg/kg.

SUMMARY:
In this study we aim to investigate the relationship between our anesthesia practice and post procedure complications after MRI scanning with sedation. This is a retrospective, single center observational study. All patients undergoing MRI scan during the study period will be included.

DETAILED DESCRIPTION:
In this study we aim to investigate the influence of patient characteristics and anesthesia choice on possible complications in patients undergoing MRI under sedation retrospectively.

After one of the routine sedation protocol used in our department was chosen and applied according to the physical status of the patient and the physicians decision, the datas of the patients will be recruited to the study from the medical records . Patient characteristics (age, gender, weight, height), ASA (American Society of Anethesiology) classification, associated diseases will be recorded . After the procedure was completed all the complications during the 2 hours waiting period in the recovery room will be recorded from the medical records. All the complşcation and recovery times will be recorded from the medical records. Whether the patient received radiocontrast material or not will also be recorded. The patients will be called by phone, and will be questioned for the complications, any epileptic seizure attack, or increase in the number of seizures, any admission to emergency room or any in patient admission to the hospital will be recorded which developed in the first week after the procedure.

ELIGIBILITY:
Inclusion Criteria:All patients undergoing MRI scan wth sedation anesthesia and giving written informed consent.

Exclusion Criteria: patients refusal to be studied.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing MRI scan wth sedation anesthesia and giving written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 977 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Patient characteristics anesthesia choice and possible complications during MRI anesthesia. | 1 week
  To investigate the influence of patient characteristics and anesthesia choice on possible complications of sedation anesthesia during MRI scanning

CONTACTS AND LOCATIONS:
Overall Officials: Ilker O Aycan, MD, Principal Investigator — Akdeniz University Hospital
Locations (1):
- AkdenizU, Antalya, Turkey (Türkiye)